CLINICAL TRIAL: NCT05538078
Title: Clinical and Radiographic Evaluation of Non-Surgical Therapy With and Without Ozone Gel Application in Controlled Type 2 Diabetic Patients With Periodontitis
Brief Title: Ozone Gel Application in Controlled Type 2 Diabetic Patients With Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Abubaker Mohamed Barahim, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ghala
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Ozone gel
  Interventions: Drug: Ozone gel
- active comparator (Active Comparator): nonsurgical periodontal treatment(scaling)
  Interventions: Drug: Ozone gel

INTERVENTIONS:
Drug: Ozone gel — application of Ozone gel after scaling by ultrasonic scaler in the bottom of periodontal pocket
  Other Names: GeliO3,Bioemmei Srl,36100 Vicenza ,Italy

SUMMARY:
The adjunctive topical subgingival application ozone gel creates a great improvements in the clinical, bacteriological and immunological parameters over the gold standard of periodontal pocket treatment alone.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of using ozone gel as a locally delivered adjunct to scaling and root planning versus scaling and root planning alone on the clinical parameters in stageIII grade B in periodontitis patients with controlled diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with controlled diabetic type II. (HgA1C <7) (Mori et al., 2021)
2. Adult patients above 18 years old.
3. Patients with stage III and grade B periodontitis.
4. Patients accept 3-months follow-up period (cooperative patients).
5. Patients provide an informed consent

Exclusion Criteria:

* 1. Presence of prosthetic crowns. 2. Extensive restorations. 3. Periodontal therapy within the last 12 months. 4. Having surgical therapy or undergoing orthodontic treatment. 5. Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis.

  6. The use of antibiotics or anti-inflammatory drugs 1 month prior to the procedure and till the end of 3 months of follow-up.

  7. Smokers. 8. Pregnant females. 9. Any known allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-08-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | 3months
  clinical attachment gain by using UNC15 Periodontal probe/ numerical data

SECONDARY OUTCOMES:
Probing Depth | 3 months
  measuring probing depth by using UNC15 Periodontal probe/numerical data
plaque index | 3 months
  measuring it visually/numerical data
Dentinal Hypersensitivity | 7 days
  measuring it using VAS scale
Bleeding on Probing visually/numerical data | 3 months
  measuring it visually/numerical data

CONTACTS AND LOCATIONS:
Overall Officials: Abeer A Barahim, BDS, Principal Investigator — Master student; Nesma M Shemais, PhD, Study Director — Lecture of oral medicine and periodontology, faculty of dentistry ,Cairo university; Mona S Darhous, PhD, Study Chair — Professor of oral medicine and periodontology factuality of Dentistry,Cairo university
Locations (1):
- Faculty of dentistry ,Cairo university, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barahim AA, Shemais N, Mousa A, Darhous M. Clinical and radiographic evaluation of non-surgical therapy with and without ozone gel application in controlled type 2 diabetic patients with periodontitis: a randomized controlled clinical trial. BMC Oral Health. 2024 Nov 25;24(1):1435. doi: 10.1186/s12903-024-05212-7. PMID 39587593